CLINICAL TRIAL: NCT03105323
Title: Role of Ratio of Progesterone to Number of Follicles as a Prognostic Tool for IntracytoplasmicSperm Injection Outcome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, ahmed nasr ali etman, Resident of Obstetrics and gynecology, Ain Shams Maternity Hospital
Other Study IDs: ain shams university
Record Dates: First submitted 2017-03-24; First posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- infertile women: All patients were pretreated with Gonadotropin releasing hormone agonist (decapeptyl®) 0.05 mg/day from 10 days prior to the start of menstruation. The patients'ovaries were stimulated with a recombinant follicle-stimulating hormone (FSH, subcutaneous) from day 2 of the menstrual cycle. human chorionic gonadotropin was administered when at least two follicles vary 18-22mm were observed on ultrasonography.Blood samples were collected on the day of final Human chorionic gonadotropin maturation, and serum P levels were measured.Pregnancy was defined by titers within 11 days following Embryo transfer,Clinical pregnancy was defined by the observation of intrauterine embryo heart motion by 7 weeks gestation.

SUMMARY:
This study will be conducted at the In vitro fertilization Unit at Ain Shams University Maternity Hospital.

Women will be recruited from the In vitro fertilization Unit who will fulfill the inclusion criteria. They will be counseled to be included into the study The study will assess Role of Ratio of Progesterone to Number of Follicles as a Prognostic Tool for Intracytoplasmic Sperm Injection outcome.

DETAILED DESCRIPTION:
Blood samples were collected on the day of final oocyte maturation, and serum Progesterone levels were measured using a chemiluminescent immunoassay for quantitative determination of the hormone .

The P/F ratio was calculated according to the equation (P(ng/mL)/number of follicles) and was defined by the measurements obtained on the day of final oocyte maturation.

All ultrasounds were performed at our In vitro fertilization center, and we included the number of follicles ≥14mm on the day of final oocyte maturation in the ratio calculation Oocytes were retrieved 36 hours after injection and were subsequently fertilized by In vitro fertilization or Intra cytoplasmic sperm injection. On day 2 - 5, all embryos were evaluated for cell number and morphology.

Each embryo transferred was evaluated for blastomere size and fragmentation. Embryos were graded as follows. Those with equal blastomere size and no fragmentation were considered Grade 1; those with blastomeres of equal size with slight fragmentation (<20 %) were Grade 2;those with blastomeres of unequal size but no fragmentation were Grade 3; those with blastomeres of equal or unequal size and moderate fragmentation (20 %-50 %) were Grade 4; and those with unrecognizable blastomeres and severe fragmentation (>50 %) were Grade 5.

The embryos were transferred on postretrieval day (2 - 5). Pregnancy was defined by Human chorionic gonadotropin titers within 11 days following Embryo transfer. Clinical pregnancy was defined by the observation of intrauterine embryo heart motion by 7 weeks gestation.

ELIGIBILITY:
Inclusion Criteria:

1. Women with any type of subfertility undergoing IVF treatment.
2. Age between (20-40) years old
3. Body mass index between (20-40)
4. Selected embryo are of grade 1 and 2 quality.

Exclusion Criteria:

1. Age above 40 years old
2. BMI above 40
3. Bad quality embryo
4. Uterine anomalies or malformation that affect embryo transfer.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: This study will be conducted at the IVF Unit at Ain Shams University Maternity Hospital.
  Women will be recruited from the IVF Unit who will fulfill the inclusion criteria. They will be counseled to be included into the study.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2017-05-01 (Estimated); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | a year
  rate of incidence of pregnancy after Intracytoplasmic Sperm Injection

IPD SHARING:
Plan to Share IPD: No